CLINICAL TRIAL: NCT02210689
Title: A Multi-center, Double-blind, Randomized Study, Comparing Clindamycin Phosphate Vaginal Cream 2% (Watson Laboratories, Inc.) to Clindesse® (Ther-Rx™, Clindamyin Phosphate Vaginal Cream 2%) and Both Active Treatments to a Placebo Control in the Treatment of Bacterial Vaginosis in Non-pregnant Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Collaborators: Watson Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-1052
Record Dates: First submitted 2014-08-04; First posted 2014-08-07 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: BACTERIAL VAGINOSIS; Signs and Symptoms to be Evaluated and Recorded Include; Vaginal Discharge Color, Odor, and Consistency; Vulvovaginal Itching and Irritation (Subjective) Absent, Mild, Moderate, or Severe; Vulvovaginal Inflammation (Objective) Absent, Mild, Moderate, or Severe
MeSH Terms: conditions — Vaginosis, Bacterial; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- test product (Experimental): One single-dose, pre-filled disposable applicator delivering approximately 5 g of cream containing approximately 100 mg of clindamycin phosphate vaginal cream 2% (Watson Laboratories, Inc.)
  Interventions: Drug: clindamycin phosphate vaginal cream 2%
- reference product (Active Comparator): One single-dose, pre-filled disposable applicator delivering approximately 5 g of cream containing approximately 100 mg of Clindesse® (clindamycin phosphate vaginal cream 2% ) (Ther-Rx™)
  Interventions: Drug: clindamycin phosphate vaginal cream 2%
- placebo (Placebo Comparator): One single-dose, pre-filled disposable applicator delivering approximately 5 g of cream containing vehicle of the test product (Watson Laboratories, Inc.)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: clindamycin phosphate vaginal cream 2%
  Arms: reference product; test product
Other: placebo — vehicle used as placebo
  Arms: placebo

SUMMARY:
A multi-center, double-blind, randomized, placebo controlled, parallel-group study, comparing Clindamycin phosphate vaginal cream 2% (Watson Laboratories, Inc.) to Clindesse® (Ther-Rx™, Clindamyin Phosphate Vaginal Cream 2%) and both active treatments to a placebo control in the treatment of bacterial vaginosis in non-pregnant women.

DETAILED DESCRIPTION:
The study treatment period will be 1 day. Subject participation is 22-30 days. Expected study duration is 10 to 12 months. The study will enroll in up to 30 clinical sites.

Test Product: One single-dose, pre-filled disposable applicator delivering approximately 5 g of cream containing approximately 100 mg of clindamycin phosphate vaginal cream 2% (Watson Laboratories, Inc.)

Reference Product: One single-dose, pre-filled disposable applicator delivering approximately 5 g of cream containing approximately 100 mg of Clindesse® (clindamycin phosphate vaginal cream 2% ) (Ther-Rx™)

Placebo Control: One single-dose, pre-filled disposable applicator delivering approximately 5 g of cream containing vehicle of the test product (Watson Laboratories, Inc.)

Dose and Mode A single applicator of investigational product cream will be administered of Administration once intravaginally at any time of the day. The subject participation is 22-30 days (drug administration for 1 day).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required study visits and must provide the written informed consent prior to any study related procedure being performed.
2. Healthy non-pregnant female aged ≥ 18 years with no known medical conditions that, in the investigator's opinion, may interfere with study participation or may interfere with the evaluation of bacterial vaginosis.
3. Female subjects of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 1 year), in addition to having a negative urine pregnancy test must be willing to use an acceptable form of birth control during the study from the day of the first dose administration to the Visit 2 Test-of-cure. For the purpose of this study the following are considered acceptable methods of birth control:

   * Oral or injectable contraceptives
   * Contraceptive patches
   * Depo-Provera® (stabilized for at least 3 months); Implanon™ (contraceptive implant), or abstinence with one of the above-listed methods of birth control should the Subject become sexually active.
   * A sterile sexual partner is NOT considered an adequate form of birth control.
   * Willing to refrain from sexual intercourse on study days 1-7 and for 48 hours prior to Visit 2 Test-of-cure.
4. Willing to refrain from using any vaginal product (e.g., spermicide, tampon, douche, diaphragm, or condom) other than study product, on study Days 1-7, for 48 hours prior to the first dose of study product, and for 48 hours prior to Visit 2 Test-of-cure.
5. Diagnosis of bacterial vaginosis, defined as the presence of all of the following:

   * Clinical diagnosis of bacterial vaginosis (e.g., thin, homogenous vaginal discharge associated with minimal or absent pruritus or inflammation AND
   * Saline wet mount of vaginal discharge demonstrating the proportion of clue cell to be ≥ 20% of the total epithelial cells AND
   * Vaginal pH > 4.5, using pH paper that measures from 4.0-6.0 AND
   * Positive "whiff test" after addition of a drop of 10% KOH to vaginal discharge)
   * Gram stain Nugent score ≥ 4 on first day of dosing (study day 1) (per Table 1 below).
   * Table 1: Nugent Scoring System (0-10) for Gram-stained Vaginal Smears (a)
   * Score (b) Lactobacillus morphotypes Gardnerella and Bacteroides spp. morphotypes Curved gram-variable rods
   * 0 4+ 0 0
   * 1 3+ 1+ 1+ or 2+
   * 2 2+ 2+ 3+ or 4+
   * 3 1+ 3+
   * 4 0 4+

Source: Nugent, R. P., M. A. Krohn, and S. L. Hillier. Reliability of diagnosing bacterial vaginosis is improved by a standardized method of Gram stain interpretation. J. Clin. Microbial. 1991; 29: 297-301.

* Morphotypes are scored as the average number seen per oil immersion field. Note that less weight is given to curved gram-variable rods. Total score = lactobacilli + G. vaginalis and Bacteroides spp/ + curved rods.
* 0, No morphotypes present; 1, <1 morphotype present; 2, 1 to 4 morphotypes present; 3, 5 to 30 morphotypes present; 4, 30 or more morphotypes present.

Exclusion Criteria:

1. Female subjects who are pregnant, nursing or planning to become pregnant during study participation.
2. Menstruating when diagnosis of bacterial vaginosis is determined at Baseline visit.
3. Primary or secondary immunodeficiency.
4. Severe liver disease.
5. History of regional enteritis, ulcerative colitis, or a history of "antibiotic-associated" colitis.
6. Evidence of any vulvovaginitis other than bacterial vaginosis. (e.g., candidiasis, Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhoeae, Herpes simplex).
7. Subjects with visible signs of HPV infection, i.e. visible warts.
8. Subject with another vaginal or vulvar condition, which would confound the interpretation of clinical response.
9. Subject will be under treatment during the study period for cervical intraepithelial neoplasia (CIN) or cervical carcinoma.
10. History of hypersensitivity to clindamycin, lincomycin, or any of the components of the vaginal creams.
11. Use within 2 weeks prior to baseline of 1) topical or systemic antibiotics or 2) topical or systemic antifungal.
12. Use of spermicides, tampons, douches, diaphragms, condoms within 48 hours of the baseline visit.
13. Concurrent use of systemic corticosteroids or systemic antibiotics.
14. Unwilling or unable to comply with the protocol requirements.
15. Subjects who have participated in an investigational drug study (i.e., subjects have been treated with an investigational drug) within 30 days prior to baseline will be excluded from study participation. Subjects who are participating in non-treatment studies such as observational studies or registry studies can be considered for inclusion.
16. Subjects who have been previously enrolled in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: nageshwar r thudi, Ph.D., CCRP, Study Director — Actavis Inc.
Locations (18):
- United States (15):
  - Akesis Investigator site 5, Birmingham, Alabama
  - Akesis Investigator site 12, La Mesa, California
  - Akesis investigator site 6, San Diego, California
  - Akesis Investigator site 1, Boynton Beach, Florida
  - Akesis investigator site 14, North Miami, Florida
  - Akesis investigator site 17, Sanford, Florida
  - Akesis investigator site 8, Sunrise, Florida
  - Akesis Investigator site 10, West Palm Beach, Florida
  - Akesis Investigator site 9, Roswell, Georgia
  - Akesis Investigator site 15, Metairie, Louisiana
  - Akesis investigator site 16, Lawrenceville, New Jersey
  - Akesis investigator site 11, Port Jefferson, New York
  - Akesis investigator site 13, Philadelphia, Pennsylvania
  - Akesis Investigator site 7, Jackson, Tennessee
  - Akesis investigator site 18, Houston, Texas
- Dominican Republic (2):
  - Akesis investigator site 3, Santo Domingo, Republica Dominicana
  - Akesis investigator site 4, Santo Domingo, Republica Dominicana
- Akesis Investigator site 2, Ponce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The populations for this study included the Safety Population, the Per-Protocol (PP) Population, and the Modified Intent-to-treat (mITT) Population.
Groups:
- Generic Clindamycin Phosphate Vaginal Cream 2%: One single-dose, pre-filled, disposable applicator of investigational product was to be administered intravaginally at home.
- Clindesse (Clindamycin Phosphate Vaginal Cream 2%): One single-dose, pre-filled, disposable applicator of Investigational product to be administered intravaginally at home.
- Vehicle Cream: One single-dose, pre-filled, disposable applicator of Investigational product was to be inserted intravaginally at home.
Period: Overall Study
Arm/Group | Generic Clindamycin Phosphate Vaginal Cream 2% | Clindesse (Clindamycin Phosphate Vaginal Cream 2%) | Vehicle Cream
Started | 242 | 240 | 122
Safety Population (Randomized participants who received the investigational product.) | 233 | 236 | 122
mITT Population (Randomized participants that applied the study dose, and returned for post-baseline evaluation visit) | 199 | 207 | 107
PP Population (Randomized subjects that were compliant with study treatment, and completed the study.) | 164 | 169 | 84
Completed | 190 | 193 | 99
Not Completed | 52 | 47 | 23
Not completed — Withdrawal by Subject | 7 | 4 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 11 | 9 | 5
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 5
Not completed — Prohibited medication | 2 | 8 | 1
Not completed — Negative Nugent score at baseline | 6 | 2 | 2
Not completed — Other | 25 | 21 | 8

BASELINE CHARACTERISTICS:
Population: Participants who received the study drug (Safety Population)
Groups:
- Clindesse (Clindamycin Phosphate Vaginal Cream 2%); Vehicle Cream: One single-dose, pre-filled, disposable applicator of investigational product was to be administered intravaginally at home.
- Total: Total of all reporting groups
Arm/Group | Generic Clindamycin Phosphate Vaginal Cream 2% | Clindesse (Clindamycin Phosphate Vaginal Cream 2%) | Vehicle Cream | Total
Number analyzed (Participants) | 233 | 236 | 122 | 591
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (9.66) | 35.8 (10.2) | 35.1 (10.17) | 35.1 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 236 | 122 | 591
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 49 | 26 | 120
  Not Hispanic or Latino | 188 | 187 | 96 | 471
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 1 | 4
  Asian | 8 | 3 | 5 | 16
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 2 | 6
  Black or African American | 94 | 106 | 55 | 255
  White | 126 | 120 | 58 | 304
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 233 | 236 | 122 | 591

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Both a Clinical and a Bacteriological Cure (Nugent Score <4), Evaluated at Visit 2 Test-of-cure (Study Day 22-30).
Description: Clinical Cure is defined as resolution of clinical signs and symptoms from entry visit as follows:
  1. The original discharge characteristic of bacterial vaginosis has returned to a normal physiological vaginal discharge which varies in appearance and consistency depending on the menstrual cycle,
  2. The whiff test is negative for any amine ("fishy") odor,
  3. The saline wet mount is negative for clue cells,
  4. Vaginal fluid pH is < 4.7, using pH paper that measures from 3.6 to 6.1.
  A Bacteriological cure is defined as a Nugent score < 4.
  The system used a 0-4 scale (Nugent Scoring System 0-10 for Gram-Stained Vaginal Smears) for evaluation of vaginal flora, based on the weighted sum of the following 3 bacterial morphotypes scores calculated from slide examination under oil immersion field:
  1. Lactobacillus: large gram positive rods,
  2. Gardnerella / Bacteroides spp: Small gram variable coccobacilli/small Gram negative rods,
  3. Mobiluncus spp.: thin, curved Gram variable rods
Time Frame: 22 to 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Test Product: One single-dose, pre-filled disposable applicator delivering approximately 5 g of cream containing approximately 100 mg of clindamycin phosphate vaginal cream 2% (Watson Laboratories, Inc.)
  clindamycin phosphate vaginal cream 2%
- Reference Product: One single-dose, pre-filled disposable applicator delivering approximately 5 g of cream containing approximately 100 mg of Clindesse® (clindamycin phosphate vaginal cream 2% ) (Ther-Rx™)
  clindamycin phosphate vaginal cream 2%
Arm/Group | Test Product | Reference Product | Placebo
Number analyzed (Participants) | 164 | 169 | 84
Participants | 36 | 34 | 9

ADVERSE EVENTS:
Time Frame: Baseline to 30 days
Description: Adverse events were collected from participants who were randomized and received the study drug.
Arm/Group | Generic Clindamycin Phosphate Vaginal Cream 2% | Clindesse (Clindamycin Phosphate Vaginal Cream 2%) | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/233 | 0/236 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/233 | 0/236 | 0/122
Other Adverse Events (participants affected / at risk) | 65/233 | 79/236 | 45/122
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Clindamycin Phosphate Vaginal Cream 2% (N=233) | Clindesse (Clindamycin Phosphate Vaginal Cream 2%) (N=236) | Vehicle Cream (N=122)
Eye Disorder (Eye disorders) | 1 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 11 | 6
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 4
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Candida infection (Infections and infestations) | 1 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 3 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 4 | 3
Oral Herpes (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 5 | 9 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Body temperature increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neoplams benign, malignant and unspecified (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Uterine leiomyoma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 2
Headache (Nervous system disorders) | 13 | 15 | 13
Migraine (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 2
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 4 | 4 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 2
Uterine spasm (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 7 | 15 | 5
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 | 3 | 1
Vaginal odour (Reproductive system and breast disorders) | 0 | 2 | 4
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 5 | 4 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 4 | 4 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 3 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 1 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 11 | 16 | 5
Vulvovaginal rash (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 | 3 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.